CLINICAL TRIAL: NCT01169012
Title: A Pharmacokinetic Study of Oral and Intravenous Clofarabine in Patients With High Risk Myelodysplasia and Acute Leukemias - Determination of Oral Bioavailability and the Effect of Cimetidine on Clofarabine Clearance
Brief Title: PK Study of Oral and IV Clofarabine in High Risk Myelodysplasia+Acute Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 0909; 10-0256 (Other: UNC OHRE)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic syndrome; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic myelomonocytic leukemia; Clofarabine; Clolar; University of North Carolina at Chapel Hill; Lineberger Comprehensive Cancer Center
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Chronic | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Trial (Other): Single Arm Trial
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Intravenous Clofarabine (10mg/m2) Oral clofarabine (30mg/m2) Cimetidine (800mg)
  Other Names: Clolar (intravenous clofarabine); Tagemet

SUMMARY:
This is a non-blinded, non-randomized pharmacokinetic study to determine the oral bioavailability of clofarabine, and the effect of cimetidine on clofarabine pharmacokinetics in patients with poor-risk acute leukemias and myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Clofarabine is a second-generation adenosine nucleoside analog with activity in hematologic malignancies. It has gained FDA-approval for use in children with relapsed-refractory ALL, and early phase studies have shown activity in patients with AML and MDS. Clofarabine's activity in acute leukemias and MDS has been established in multiple phase I and II studies, both alone and in combination with cytosine arabinoside (araC), and in both relapsed-refractory patients, and untreated older adults.

Pharmacokinetic investigations comparing I.V. and P.O. dosing within the same patient have not been performed. Furthermore, the effect of OCT2 inhibition on clofarabine pharmacokinetics in humans has not been investigated. The potential for enhanced drug exposure and toxicity in the setting of OCT2 inhibition is of clinical importance as clofarabine gains broader indications in hematologic oncology. In particular, bioavailability and the OCT2 mechanism are important with prolonged drug exposure and oral administration in older adults, who are likely to have impaired renal function and take other drugs that interact with OCT2 such as metformin (a substrate) and trimethoprim (one of several inhibitors). OCT2 is expressed on several solid tumor cell lines, and is thought to play a role in tumor uptake of cationic cytotoxins. Whether OCT2 or other transporters are expressed on leukemic blasts, or influence drug uptake has not been investigated. However, variation in the expression of drug transporters could be one of several mechanistic explanations for the fact that clofarabine-responsive patients accumulate intracellular clofarabine triphosphate, whereas non-responders do not.

Single nucleotide polymorphisms have been identified in the gene encoding OCT2, which may influence substrate uptake or inhibitor potency. Such polymorphisms may explain variation in clofarabine pharmacokinetics and pharmacodynamics between individuals, but the potential for this phenomenon has not previously been investigated.

Patients will receive clofarabine as induction therapy in five doses. Initially, and unless dose escalation or de-escalation criteria are met, patients will be assigned to dose level 0 (IV Clofarabine 15mg/m2; Oral clofarabine 30mg/m2). The first three doses (on days 1, 3 and 5) will be administered followed by washout periods that extend until the next clofarabine dose is administered. During the washout periods, frequent phlebotomy for PK sampling will be performed in an outpatient setting at the UNC Clinical Translational Research Center (CTRC). The duration of the induction period will be determined by time to recovery of hematologic toxicity (platelets >50 x 109/liter, ANC >1.0x109/liter).

AML patients achieving CR, and MDS patients achieving CR, PR or hematologic improvement will receive additional consolidation cycles of oral clofarabine daily on days 1 through 5 of each subsequent cycle, with clofarabine dose according to assigned dose level (0: 30 mg/m2, -1: 20 mg/m2, +1: 40 mg/m2). Consolidation cycles will begin no sooner than 28 days after the first day of the previous clofarabine cycle. Patients will be evaluated for response after each cycle, and will be continued on trial for up to 6 total cycles of therapy as long as a response or lack of progression is maintained and no Grade 3-4 non-hematologic toxicities have been observed in that patient.

ELIGIBILITY:
Inclusion Criteria:

* MDS patients age 18 and older with IPSS risk of intermediate-2 who have failed ≥ 1 prior regimen with a DNA methyltransferase inhibitor, or have ≥ 10% bone marrow myeloblasts
* MDS patients age 18 and older with IPSS high risk
* Patients with CMML (chronic myelomonocytic leukemia) age 18 and older
* Untreated AML or Ph-negative ALL patients age 60 and over who are deemed not to be candidates for intensive anthracycline based induction therapies based on age, organ function or co-morbidities
* AML or Ph-negative ALL patients age 60 and over who have failed or relapsed following initial induction therapy
* Provide signed written informed consent.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Serum creatinine </= 1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min as calculated by the Cockcroft-Gault equation:

GFR (mL/min) = (140 - age) X (weight in kg) X (0.85 if female)/ 72 X serum creatinine in mg/mL

* Serum bilirubin ≤1.5 mg/dL × upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) </=2.5 × ULN
* Alkaline phosphatase 2.5 × ULN

  * Female patients of childbearing potential must have a negative serum pregnancy test within 1 week prior to enrollment.
  * Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
  * INR ≤ 1.5 and APTT within the upper limits of normal (Patients on therapeutic anticoagulation will be allowed to participate if anticoagulation can be changed to parenteral medication or discontinued when platelet count is <50x109/liter)

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Abnormal organ function as defined by ALT, AST or total bilirubin >1.5 x ULN, GFR< 60mL/minute by MDRD equation
* Active cardiac disease as manifest by: >class II NYHA congestive heart failure, unstable angina or myocardial infarction within the last 6 months
* Hemorrhage or bleeding >/= CTCAE grade 3 within 4 weeks of enrollment
* Pulmonary hemorrhage >/= CTCAE grade 2 within 4 weeks of enrollment
* HIV infection
* Active Hepatitis B or Hepatitis C infection (defined as measurable viral load by PCR, or liver function abnormalities attributed to viral hepatitis)
* Cerebrovascular accident or transient ischemic attack within 6 months of study enrollment.
* Non-healing wound or ulcer, or major surgery or trauma within 4 weeks of study enrollment
* Active graft versus host disease of any grade
* Active CNS disease that will require radiation therapy.
* Suspected or confirmed hypersensitivity to cimetidine or other histamine H2 antagonists.
* Have currently active gastrointestinal disease, or prior surgery that may affect the ability of the patient to absorb oral clofarabine.
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Medical indication for therapy with one of the previously-documented human OCT2 inhibitors (table 4), for which cessation of the OCT2 inhibitor or conversion to an alternate agent would pose unacceptable risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Define human intra-patient bioavailability of clofarabine; Compare the pharmacokinetics of intravenously-administered clofarabine when administered alone, with the pharmacokinetics of clofarabine when co-administered with cimetidine, an OCT2 inhibitor. | 4 years
  Regarding primary endpoints, each patient will generate pharmacokinetic data sufficient to compute area under the concentration versus time curve (AUC) and clearance (Cl) for each of the initial three clofarabine doses (IV, PO and IV administered after cimetidine) for each patient.
  These values will be used to compute the human oral bioavailability of clofarabine and compare AUC and Cl of clofarabine when given after cimetidine with AUC and Cl of clofarabine when administered alone

SECONDARY OUTCOMES:
Examine safety of orally-administered clofarabine; Examine the safety of a combined intravenous and oral clofarabine regimen | 5 Years
  Regarding secondary objectives, safety will be evaluated by grading and reporting all adverse experiences during protocol therapy.
  The DLT rate of ≤ 20% is considered to be acceptable.
Examine efficacy of orally-administered clofarabine | 5 years
  Response to therapy will be determined at the time of hematologic reconstitution (platelets >50 x 109/liter, ANC >1.0x109/liter for MDS patients or platelets >100 x 109/liter, ANC >1.0x109/liter for leukemia patients) or day 28, whichever is sooner by complete blood count with differential and bone marrow aspirate, biopsy and cytogenetics.
Explore the influence of OCT2-encoding single nucleotide polymorphisms on clofarabine pharmacokinetics and pharmacodynamics | 5 years
  The effect of previously-described OCT2 polymorphisms on clofarabine pharmacokinetics will be investigated in an exploratory study. If specific OCT2-encoding single nucleotide polymorphisms are detected in study subjects, the geometric mean AUC and Cl of clofarabine in such patients will be compared with the geometric mean AUC and Cl in patients with wild-type OCT2.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Foster, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center Home Page — http://unclineberger.org/
- See also: Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials